CLINICAL TRIAL: NCT05648045
Title: Associations Between Factors Contributing to Obesity (Dietary Behaviour and Physical Activity), Resilience (Dietary and Physical Activity Self-Efficacy, Self- Esteem, General Resilience and Optimism), and HRQoL in Indian Adolescents
Brief Title: Resilience and Obesity Prevention in Adolescents
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: Resilient Kids
Record Dates: First submitted 2022-11-22; First posted 2022-12-13 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Obesity, Childhood; Self Efficacy; Optimism; Resilience, Psychological; Quality of Life; Self Esteem
Keywords: psychosocial resilience; obesity prevention; adolescents; quality of life; weight resilience
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Groups classified based on BMI: Group 1: Overweight BMI Cut-Off Points (kg/m²) by International Obesity Task Force; IOTF Overweight (including obesity) ≥25.00
  Group 2: Obese BMI Cut-Off Points (kg/m²) by International Obesity Task Force; IOTF
  Obese ≥30.00
  Group 3: Normal-weight BMI Cut-Off Points (kg/m²) by International Obesity Task Force; IOTF
  Healthy Weight - 18.5-24.99

SUMMARY:
A cross-sectional observation study to see the associations between factors contributing to obesity , resilience, and HRQoL in Indian adolescents.

Study objectives :

1. To classify consenting adolescents into normal, underweight, overweight, and obese groups.
2. To assess diet and physical activity self-efficacy, self-esteem, general resilience, optimism, and HRQoL in the above groups.
3. To compare the differences in the groups between factors contributing to obesity (dietary behavior and physical activity), resilience (diet and physical activity self-efficacy, self-esteem, general resilience, and optimism), and HRQoL in Indian adolescents

Main research question:

Is there a relationship between resilience (measured as diet and physical activity self-efficacy, self-esteem, general resilience, and optimism) and BMI Z score in 14 - 16 years old school children from Kolkata?

To answer this, the following sub-questions will be studied:

1. Is there a difference in resilience between the different groups of children (underweight, normal, overweight and obese)? To investigate this question, the level of diet and physical exercise self-efficacy, self-esteem, general resilience, and optimism will be investigated among overweight, obese, underweight, and normal-weight adolescents while controlling for age, gender, and type of school.
2. Is there a relationship between HRQoL and BMI Z score in different groups of children (underweight, normal, overweight and obese)? To investigate this question, the level of HRQoL will be investigated among overweight, obese, underweight, and normal-weight adolescents while controlling for age, gender, and type of school.
3. Is there a relationship between resilience and dietary behavior and physical activity in different groups of children (underweight, normal, overweight and obese) controlling for age, gender, socio-economic status and type of school?
4. Is there a relationship between parents' nutrition knowledge and resilience in children? To investigate this question, the level of parents' nutrition knowledge will be investigated among underweight, normal, overweight and obese adolescents while controlling for age, gender, and type of school.

DETAILED DESCRIPTION:
Childhood obesity is associated with increased health risks in adulthood, affecting capacity for physical activity and occupational performance, as well as psychological and social deficits. These are significant contributors to direct and indirect costs. The prevalence of obesity and related factors in young children emphasizes the importance of understanding periods of vulnerability in early development and the interaction between physical activity, lifestyle, and dietary behaviour, resilience, and HRQoL. Factors for preventing obesity are social support and a person's willingness to lifestyle changes (Gilchrist & Zametkin, 2006). With many adverse effects of adolescent obesity, one's resilience (self-esteem, self-efficacy, and optimism) may contribute to being protective, ultimately influencing the individual's overall health-related quality of life. However, to the investigator's knowledge, resilience (self-esteem, self-efficacy, and optimism) has not been explored from the perspective of a protective factor to obesity development, particularly in Indian adolescents.

The study aims to identify the relationship between resilience and obesity factors in Indian adolescents. The main aim of this study is to see the correlation of resilience, identified as self-esteem, diet and physical exercise self-efficacy, and optimism, with factors influencing the development of obesity (physical activity, lifestyle, and dietary behaviour) in Indian children/adolescents. In this cross-sectional study, samples will be recruited from sites where other influencing factors can be controlled, for example the local secondary schools (where investigators can control for socioeconomic background, education, etc.)

The current study findings may lead to a holistic understanding of obesity-contributing factors, such as dietary habits and physical activity and their relationship with resilience and HRQoL. Increased knowledge of these factors may lead to more comprehensive studies involving resilience and obesity and also study if the early resilience-building intervention can potentially lower the chances of developing obesity in adolescents. Results from the study can also help build more effective programs for health professionals and nutritionists striving to reduce or prevent obesity among adolescents. Results from the present study maybe used by future researchers to develop interventions to strengthen resilience among children at risk for overweight or obesity.

Process for participant recruitment process in India: Schools will be selected through previously established professional networks of the student researcher. A snowball or chain sampling strategy will be followed to recruit the schools. In this form of recruitment, selected participants identify other potential informants. Through snowballing (Kaplan et al., 1987), school principals previously known to the student researcher will help to identify other school principals as potential participants for the study. This will be followed by face-to-face meetings with the principals of identified schools, and they will be requested to participate in the study after explaining the details. The school principal will facilitate the recruitment of students and parents. The number of schools chosen will depend on the total sample size for the study. Both private and government schools will be selected. After completing the school selection, the researcher will visit each school and meet the school principal to brief about the research study. Participation in the study is voluntary. School involvement will be minimal. A detailed study brochure will be handed over to the school principal for uploading to the school notice board. The school principal will facilitate the recruitment of students and share the study details through an announcement in the school assembly. Parent questionnaires and consent forms will be sent home with the child. Once the parent agrees to participate in the study, they can send the signed consent and filled-out questionnaires with the student to school. The student needs to submit it to the concerned person in school from where the researcher will collect it back. The researcher will briefly explain the study to the class teacher and the students through a one-time meeting. Data collection for children will happen during school recess/after school.

The study will have two phases: a pilot phase and a main phase. The findings from the pilot will help determine the questionnaire design for the main phase.

ELIGIBILITY:
Inclusion Criteria:

* Children who are underweight, overweight, children with obesity, and children with normal body weight based on IOTF cut-offs
* otherwise healthy, without any confirmed diagnosed clinical/mental illness
* age between 14-16 years
* agreed to participate

Exclusion Criteria:

* confirmed diagnosed clinical/mental illness
* more than 16 years, less than 14 years of age

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Indian children who are underweight, overweight, obese, and normal weight according to the International Obesity Task Force (IOTF) criteria
  Otherwise healthy, without any confirmed diagnosed clinical/mental illness, aged between 14-16 years
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Outcome = resilience (numerical variable) Main determinant = normal weight versus overweight/obese (binary) | At 1 year
  Total score measured for each of the following: diet and physical activity self-efficacy, self-esteem, general resilience, and optimism

SECONDARY OUTCOMES:
Health-related quality of life (HRQOL) | At 1 year
  Total score measured for Pediatrics Quality of Life: PedsQL

CONTACTS AND LOCATIONS:
Overall Officials: Poulami Dasgupta, Principal Investigator — Maastricht University/MaastrichtUMC
Locations (16):
- India (16):
  - Mitra Institution (Main), Kolkata, West Bengal
  - Victoria Institution High School, Kolkata, West Bengal
  - Ballygunge Government High School, Kolkata, West Bengal
  - Andhra Association High School (AAHS), Kolkata, West Bengal
  - Lycee School, Kolkata, West Bengal
  - National High School For Boys, Kolkata, West Bengal
  - National High School For Girls, Kolkata, West Bengal
  - Tollygunge Adarsh Hindi High School (Girls and Boys), Kolkata, West Bengal
  - New Alipore Multipurpose School, Kolkata, West Bengal
  - New Vista Academy, Kolkata, West Bengal
  - Sakhawat Memorial Govt. Girls' High School, Kolkata, West Bengal
  - Calcutta Public School, Bidhan Park, Kolkata, West Bengal
  - Indus Valley World School, Kolkata, West Bengal
  - Calcutta Public School, Kalikapur, Kolkata, West Bengal
  - Holy Mission school, Kolkata, West Bengal
  - St. Joseph and Mary's school, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Undecided